CLINICAL TRIAL: NCT06937775
Title: Rapid Maxillary Expansion Related Sutural and Dentoalveolar Changes Provoke Salivary Oxidative Stress: A Biochemical Study
Brief Title: Rapid Maxillary Expansion Related Oxidative Stress and Periodontal Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek KARADOĞAN, Assoc. Prof. Dr., Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: BAP 2015/306
Record Dates: First submitted 2025-03-29; First posted 2025-04-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-04

CONDITIONS: Maxillary Expansion
MeSH Terms: interventions — Dental Plaque Index; Periodontal Index

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- TO (Other): 1 week before the placement of the Hyrax appliance
  Interventions: Other: Periodontal measurements (plaque index, gingival index and probing pocket depth scores ); Other: Biochemical Sample Supply (Collection of serum and saliva samples)
- T1 (Other): The day of the first clinical observation of sutural opening (5-7 days after activation)
  Interventions: Other: Periodontal measurements (plaque index, gingival index and probing pocket depth scores ); Other: Biochemical Sample Supply (Collection of serum and saliva samples); Procedure: Rapid maxillary expansion with Hyrax appliance
- T2 (Other): The day of completion of active expansion (3-4 weeks)
  Interventions: Other: Periodontal measurements (plaque index, gingival index and probing pocket depth scores ); Other: Biochemical Sample Supply (Collection of serum and saliva samples); Procedure: Rapid maxillary expansion with Hyrax appliance
- T3 (Other): The day of completion of the 3-month reinforcement period
  Interventions: Other: Periodontal measurements (plaque index, gingival index and probing pocket depth scores ); Other: Biochemical Sample Supply (Collection of serum and saliva samples); Procedure: Rapid maxillary expansion with Hyrax appliance

INTERVENTIONS:
Other: Periodontal measurements (plaque index, gingival index and probing pocket depth scores ) — Plaque index (PI), gingival index (GI) and probed pocket depth (PPD) scores will be recorded at T0, T1, T2 and T3 assessment periods to evaluate the periodontal status and oral care effectiveness of the participants. PPD is the distance between the gingival margin and the sulcus base. Measurements will be made at 6 different sites (mesio-vestibular, vestibular, disto-vestibular, mesio-oral, oral, disto-oral) of each tooth using a Williams periodontal probe (Hu Friedy, Chicago, Illinois, USA). During the measurements, care will be taken to position the probe as parallel as possible to the long axis of the tooth and not to apply excessive force.
Other: Biochemical Sample Supply (Collection of serum and saliva samples) — Serum and saliva samples will obtained from all individuals included in the study at T0, T1, T2 and T3 for biochemical analyses.
  For standardisation purposes, blood samples will be collected from the antecubital fossa with the patients in a sitting position. After resting for 30 minutes (min) at room temperature, the samples will be centrifuged (4ºC at 3000 rpm for 5 min) and serum samples will be obtained. The samples will be transferred into eppendorf tubes and stored in the freezer (-80ºC) until the study day.
  Sampling will be performed early in the morning. Participants will be warned not to consume anything other than water for the last 12 hours and not to brush their teeth that morning. Individuals will be left with their mouths open for 5 min to allow saliva to accumulate at the floor of the mouth. Unstimulated saliva samples accumulated at the floor of the mouth will be collected and transferred to eppendorf tubes.
Procedure: Rapid maxillary expansion with Hyrax appliance — Rapid maxillary expansion (RME) is the most commonly preferred treatment of skeletal jaw stenosis in the transversal direction. Bilateral anchorage is the process of increasing the transversal dimension of the midpalatal suture (sutura palatina media) by applying strong tensile forces in the lateral direction to the dentoalveolar structures of the teeth and/or palatal bone. The primary goal of treatment is to provide orthopedic movement through sutural separation.
  Arms: T1; T2; T3

SUMMARY:
The aim of this study was to investigate the effects of rapid maxillary expansion on local and systemic oxidative stress levels. Thirty-five volunteer patients (17 females and 18 males) who needed rapid maxillary expansion will be included in the study. Serum and saliva samples will be collected from each patient during four different periods: a week before the treatment (T0), on the day of sutural separation (T1), at the end of the active expansion period (T2), and after the completion of a 3-month retention period (T3). To evaluate the patients' periodontal status, plaque index, gingival index, and probing pocket depth scores will be recorded for each period. 8-hydroxydeoxyguanosine (8-OHdG), total oxidative status (TOS), total antioxidant capacity (TAS), and oxidative stress index (OSI) biomarkers will be evaluated to determine the local and systemic oxidative stress levels.

ELIGIBILITY:
Inclusion Criteria:

* Being between 11-15 years of age,
* Having an indication for maxillary expansion due to maxillary stenosis,
* Being highly cooperative, performing adequate oral care,
* Being periodontally healthy,
* Not having cleft lip and/or palate anomalies,
* Not having any systemic disease,
* Not having used any medication including antibiotics and anti-inflammatory drugs in the last 6 months,
* Not being substance addicted and not smoking.

Exclusion Criteria:

* Having inadequate oral hygiene
* Being periodontally unhealthy
* Having cleft lip and/or palate anomalies,
* Having any systemic disease,
* Having used any medication including antibiotics and anti-inflammatory drugs in the last 6 months,
* Being substance addicted and not smoking.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2016-01-10 (Actual); Primary Completion 2016-03-10 (Actual); Study Completion 2016-08-10 (Actual)

PRIMARY OUTCOMES:
Biochemical analyses - 8-OHdG | a week before the treatment (T0), 5-7 days after activation (T1), 3rd week (T2), and after the completion of a 3-month retention period (T3)
  8-OHdG is the most frequently encountered and best known mutagenicity of more than 20 oxidative base damage products of ROS in DNA. Since it is easily detected in living cells and body fluids, it is the most commonly used oxidative DNA damage marker.
  Serum and saliva levels will be measured using a suitable ELISA kit (Cayman Chemical DNA/RNA Oxidative Damage ELISA Kit Item No.589320) according to the manufacturer's instructions. The measurement principle is as follows: It is based on the competition between 8-OHdG from the sample and 8-OHdG-acetylcholinestarase conjugate (8- OHdG Tracer) from the kit for a limited amount of 8-OHdG monoclonal antibody covering the plate well. The colour intensity measured spectrophotometrically at 410 nm is directly proportional to the tracer and inversely proportional to the amount of free 8-OHdG in the sample.
Biochemical analyses - Oxidative Stress Index (TOS/TAS=OSI) | a week before the treatment (T0), 5-7 days after activation (T1), 3rd week (T2), and after the completion of a 3-month retention period (T3)
  Total Oxidative Status (TOS) is a current method used to detect lipid peroxidation and oxidative stress. TOS is considered to be a superior method compared to other methods due to the impracticality of measuring different oxidant molecules individually and the inability to fully reflect the interaction of oxidant molecules with each other. Total Antioxidan Status (TAS) is a biochemical parameter obtained as a result of the sum of the antioxidant capacities of all antioxidants in the biological samples examined. Oxidative Stress Index (OSI) is a proportional value obtained by dividing TOS by TAS. It is directly affected by total oxidative and antioxidant status and reveals the final oxidative status in a practical and understandable way.
  OSI value was calculated according to the following formula. OSI = TOS (mmol H2O2 Equiv./L) / TAS (mmol Trolox Equiv./L) x 100

SECONDARY OUTCOMES:
Clinical Periodontal Assessments-plaque index | a week before the treatment (T0), 5-7 days after activation (T1), 3rd week (T2), and after the completion of a 3-month retention period (T3)
  Plaque index (PI) scores will be recorded at T0, T1, T2 and T3 assessment periods to evaluate the periodontal status and oral care effectiveness of the participants. The amount and thickness of plaque causing gingival inflammation will be determined. The teeth will be dried by spraying light air and isolated. Each tooth will be scored by measuring with a probe from the gingival margin in six areas (mesiobuccal, distobuccal, mesial, distal, oral, vestibule).
Clinical Periodontal Assessments-gingival index | a week before the treatment (T0), 5-7 days after activation (T1), 3rd week (T2), and after the completion of a 3-month retention period (T3)
  Gingival index (GI) scores will be recorded at T0, T1, T2 and T3 assessment periods to evaluate the periodontal status of the participants. The periodontal probe will be placed in the gingival sulcus parallel to the long axis of the teeth from the gum edge. Measurements will be made from the area under the teeth and scoring will be done according to the surface characteristics of the gum. The value found will be divided by the number of teeth and the gingival index will be determined for the entire mouth.
Clinical Periodontal Assessments-probed pocket depth (PPD) | a week before the treatment (T0), 5-7 days after activation (T1), 3rd week (T2), and after the completion of a 3-month retention period (T3)
  PPD is the distance between the gingival margin and the sulcus base. Measurements will be made at 6 different sites (mesio-vestibular, vestibular, disto-vestibular, mesio-oral, oral, disto-oral) of each tooth using a Williams periodontal probe (Hu Friedy, Chicago, Illinois, USA). During the measurements, care will be taken to position the probe as parallel as possible to the long axis of the tooth and not to apply excessive force.